CLINICAL TRIAL: NCT05775614
Title: Study of Uro-Tainer® Polihexanide and Uro-Tainer® With Citric Acid on Catheter Blockage, Infection Prevention, Cost-effectiveness and Quality of Life (UROBIQ): a Prospective Randomized Single-blinded Clinical Study
Brief Title: UROtainer for Bladder Catheter Maintenance, Infection Prevention and Quality of Life
Acronym: UROBIQ
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Karin Andersen, Principal Investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UROBIQ
Record Dates: First submitted 2022-12-17; First posted 2023-03-20 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Catheter Blockage
Keywords: Catheter maintenance; UroTainer; prophylactic; catheter flushing

STUDY DESIGN:
Intervention Model Description: 2 arms with randomization 1:1
  1. Uro-Tainer® Polihexanide two weekly rinses compared to two weekly rinses with saline for 3 months.
  2. Uro-Tainer® with citric acid: Two weekly rinses compared to two weekly rinses with saline for 3 months.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Uro-Tainer® catheter flushing (Experimental): Uro-Tainer® catheter flushing two times weekly for 3 months.
  Interventions: Device: UroTainer®
- Saline catheter flushing (Placebo Comparator): Saline solution catheter flushing two times weekly for 3 months.
  Interventions: Device: Saline

INTERVENTIONS:
Device: UroTainer® — Clinical effect of preventive treatment - catheter flushing with UroTainer®
  Arms: Uro-Tainer® catheter flushing
Device: Saline — Clinical effect of preventive treatment - catheter flushing with saline solution
  Arms: Saline catheter flushing

SUMMARY:
The purpose of the current study is to investigate whether catheter flushing with Uro-Tainer® with citric acid and Uro-Tainer® Polihexanide can: Reduce catheter changes due to incrustation and blockage.

In addition, a list of secondary aims inclusive of cost-effectiveness analysis in collaboration with the Centre for Innovative Medical Technology (CIMT) at OUH.

DETAILED DESCRIPTION:
The purpose of the current study is to investigate whether catheter flushing with Uro-Tainer® with citric acid and Uro-Tainer® Polihexanide can: Reduce catheter changes due to incrustation and blockage.

In addition, a list of secondary aims inclusive of cost-effectiveness analysis in collaboration with the Centre for Innovative Medical Technology (CIMT) at OUH.

There is a need for a randomised study to justify if Uro-Tainer® flushing will have an advantage over the cheaper and normally used Saline flushing.

Standard therapies vary depending on the blockage type and severity. Saline Solution can be used daily for a shorter period and 1-2 times a week for long-term catheter maintenance.

Study:

* Uro-Tainer® Polihexanide two weekly rinses compared to two weekly rinses with saline for 3 months.
* Uro-Tainer® with citric acid: Two weekly rinses compared to two weekly rinses with saline for 3 months.

Clinical benefits:

* Less catheter blockage -> less need for catheter replacement outside the regular schedule -> Fewer infections and better QoL
* It is expected that cost-effectiveness analysis will show a better economic outcome for the society
* No unknown adverse effects are expected
* The risk of participation in this study is very small compared to the expected effect of fewer catheter replacements, fewer infections and better QoL which justifies the selection of clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

Citizen not previously flushed

* A permanent catheter (suprapubic and urethral)
* Male and female > 18 years of age
* Acute or previous catheter stop because of blocking or incrustations.
* The pilot project does not include clogging due to incrustations
* Voluntary consent to participate in the study, following a full explanation of the nature and purpose of the study, by signing the informed consent form approved by the Ethics Committee (EC) before all evaluations.

Citizen previously flushed with NaCl or UroTainer®

* A permanent catheter (suprapubic and urethral)
* Male and female > 18 years of age
* Willingness to take a rinse break for a minimum of 4 weeks. In the event of 2 catheter stops during the flushing break, assessed on the basis of an urgent need for catheter flushing with NaCl or catheter change, the citizen can be included.
* The pilot project does not include clogging due to incrustations
* If there is no catheter stop during the rinsing break, the citizen will continue without rinsing until a possible catheter stop.
* Voluntary consent to participate in the study, following a full explanation of the nature and purpose of the study, by signing the informed consent form approved by the Ethics Committee (EC) before all evaluations.

Exclusion Criteria:

* Urothelial cancer
* Bladder and kidney stones requiring treatment
* Age < 18 years of age
* Pregnant and / or breastfeeding women
* Not able to understand Danish
* Dementia, where relatives can / will not give consent
* Simultaneous participation in another interventional clinical trial (drugs or medical devices studies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of catheter changes during the treatment and follow-up period. | 1 year
  Number of catheter changes

SECONDARY OUTCOMES:
UTI events (Urinary tract infection event) | 1 year
  The number of prescriptions
Urine culture | 1 year
  Urine culture performed if UTI is suspected
Odour | 1 year
  Odour nuisance is to be assessed on a 5-point scale. A high score is a worse outcome.
  1. No odour
  2. Discreet odour nuisance after catheter care
  3. Odour that is noticed once in a while. Noticed by the participant and relatives
  4. Odour that is present all the time around the participant
  5. Solid odour that is felt in all rooms. "It hangs" on the participant
Quality of life by SF-36 | 1 year
  SF-36 (Health Survey Short Form 36)
  The SF-36 consists of 36 items - that are grouped into 8 subscales or domains:
  Physical functioning (10 items); Role limitations due to physical health (4 items); Role limitations due to emotional problems (4 items); Energy/fatigue; Emotional well-being; Social functioning (2 items); Pain (2 items); General health. Aggregate scores for each domain range from 0 to 100, compiled as a percentage - where the higher the score, the more favourable the health state.
Quality of life by ICIQ-LTCqol | 1 year
  Living with a long term catheter (ICIQ-LTCqol 12/12 ) The questionnaire consists of three scales yielding two summary measures catheter function and concern score, lifestyle impact and unscored items. Possible scores range from 1 to 530, with lower scores representing better catheter function, concern score and life impact.
Cost effectiveness analyses 1 | 1 year
  Costs of used catheters in DDK pr participant
Cost effectiveness analyses 2 | 1 year
  Costs of used solutions for the maintenance of indwelling urethral and suprapubic catheters in DKK pr participant
Cost effectiveness analyses 3 | 1 year
  Costs of used time of the health care professionals used for catheter maintenance and control in primary care in DKK pr participant

CONTACTS AND LOCATIONS:
Overall Officials: Karin Andersen, Principal Investigator — University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No